CLINICAL TRIAL: NCT01903070
Title: EFFECTS OF LINAGLIPTIN ON ACTIVE GLP-1 CONCENTRATIONS IN SUBJECTS WITH RENAL IMPAIRMENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00/0594-LINARI
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin in TD2 subjects (Experimental): Linagliptin in TD2 subjects with normal renal function
  Interventions: Drug: Linagliptin
- Linagliptin in TD2 subjects with impaired renal function (Experimental): Linagliptin in TD2 subjects with impaired renal function
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin

SUMMARY:
This is a bi-centric, prospective, open study comparing the effects of linagliptin on active GLP-1 concentrations in subjects with renal impairment compared to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 diabetes mellitus based on the disease diagnostic criteria (WHO) classification

Exclusion Criteria:

* Subjects with type 1 diabetes, maturity onset diabetes of the young (MODY) or secondary forms of diabetes such as due to pancreatitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
ΔAUCGLP-1-OGTT(0-240) | Glucose tolerance test following 7 days of therapy
  ΔAUCGLP-1-OGTT(0-240) Change in active GLP-1 concentrations after oral glucose ingestion after linagliptin Treatment compared between Groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany